CLINICAL TRIAL: NCT00390104
Title: Molecular Analysis of Nucleic Acids Derived From Patients With Neuromuscular Disease and Their Family Members
Brief Title: Molecular Analysis of Patients With Neuromuscular Disease
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Louis Kunkel, Professor of Genetics and Pediatrics, Harvard Medical School, Boston Children's Hospital
Other Study IDs: 03-12-205; 5R01NS080929 (NIH)
Record Dates: First submitted 2006-10-17; First posted 2006-10-19 (Estimated); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Neuromuscular; Disorder, Hereditary; Duchenne/Becker Muscular Dystrophy; Limb-girdle Muscular Dystrophy
Keywords: Neuromuscular Disease; Muscle weakness; Muscle atrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Dystrophies, Limb-Girdle; Neuromuscular Diseases; Muscle Weakness; Muscular Atrophy

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from blood or saliva from proband, Muscle tissue from proband, DNA from blood or saliva from family members, Skin biopsy from proband and family members
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to identify new genes responsible for neuromuscular disorders and study muscle tissue of patient with known neuromuscular disease, as well as their family members. We are interested in recruiting many types of neuromuscular disease including; Duchenne muscular dystrophy (DMD), Becker muscular dystrophy (BMD), and limb-girdle muscle dystrophy (LGMD). There are still many patients diagnosed with muscular dystrophy with no causative gene implicated in their disease. Using molecular genetics to unravel basis of these neuromuscular disorders will lead to more accurate diagnosis/prognosis of these disorders which will lead to potential therapies.

DETAILED DESCRIPTION:
We are looking to discover new disease genes responsible for the neuromuscular diseases found in our participants and their families. Our research lab has a long history of identifying novel genes responsible for various forms of neuromuscular disease including; DMD gene, the sarcoglycans, obscurin, and filamin. Each discovery has resulted in advances in our ability to develop diagnostic tests which benefit patients and their families by providing accurate diagnosis, presymptomatic and/or prenatal testing. Genotype-phenotype correlation studies have increased our understanding of the natural history of these rare disorders benefiting patients through better prognostic determinations by clinicians. Biochemical and pathological analysis of muscle biopsy samples in patients with known and unknown types of neuromuscular disease has led to new insights into disease pathophysiology, which we hope will aid in finding new treatments.

ELIGIBILITY:
The samples used in this study will be derived from individuals at risk for, or suffering from, neuromuscular disease, generally resulting in clinical weakness of one or more muscle groups and their family members.

Inclusion criteria:

1. having a clinical and/or pathological diagnosis of a muscular dystrophy
2. being the first degree relative of someone with such a diagnosis
3. having had a muscle biopsy if diagnosed with a neuromuscular disease
4. willingness to provide a skin biopsy for research only

Exclusion Criteria:

1. not having a neuromuscular diagnosis in you or a family member
2. not wishing to participate
3. being incapable of giving consent and not having a legal guardian willing or able to do so

Ages: 1 Week to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Families will be ascertained world-wide as the muscular dystrophies are a pan-ethinic group of diseases.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2002-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Louis M Kunkel, PhD, Principal Investigator — Boston Children's Hospital/Harvard Medical School
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be de-identified to protect privacy, but maybe shared with other researchers.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Once a participant is enrolled, we will keep the data indefinitely.
Access Criteria: Data will only be shared with collaborating scientists once a patient enrolls. Data will be shared according to choice on individual consent forms.

REFERENCES:
- [Background] Saha M, Reddy HM, Salih MA, Estrella E, Jones MD, Mitsuhashi S, Cho KA, Suzuki-Hatano S, Rizzo SA, Hamad MH, Mukhtar MM, Hamed AA, Elseed MA, Lek M, Valkanas E, MacArthur DG, Kunkel LM, Pacak CA, Draper I, Kang PB. Impact of PYROXD1 deficiency on cellular respiration and correlations with genetic analyses of limb-girdle muscular dystrophy in Saudi Arabia and Sudan. Physiol Genomics. 2018 Nov 1;50(11):929-939. doi: 10.1152/physiolgenomics.00036.2018. Epub 2018 Aug 31. PMID 30345904
- [Result] Vieira NM, Spinazzola JM, Alexander MS, Moreira YB, Kawahara G, Gibbs DE, Mead LC, Verjovski-Almeida S, Zatz M, Kunkel LM. Repression of phosphatidylinositol transfer protein alpha ameliorates the pathology of Duchenne muscular dystrophy. Proc Natl Acad Sci U S A. 2017 Jun 6;114(23):6080-6085. doi: 10.1073/pnas.1703556114. Epub 2017 May 22. PMID 28533404
- [Result] Reddy HM, Cho KA, Lek M, Estrella E, Valkanas E, Jones MD, Mitsuhashi S, Darras BT, Amato AA, Lidov HG, Brownstein CA, Margulies DM, Yu TW, Salih MA, Kunkel LM, MacArthur DG, Kang PB. The sensitivity of exome sequencing in identifying pathogenic mutations for LGMD in the United States. J Hum Genet. 2017 Feb;62(2):243-252. doi: 10.1038/jhg.2016.116. Epub 2016 Oct 6. PMID 27708273